CLINICAL TRIAL: NCT02360566
Title: The Novel Use of Participatory Video as a Recovery-Oriented Intervention in Early Psychosis: A Pilot Study
Brief Title: Participatory Video as a Recovery-Oriented Intervention in Early Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: ProjectVideo Inc. (Industry); London Health Sciences Centre (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Arlene MacDougall, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8211
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: Psychosis; Schizophrenia; Participatory Video; Narrative
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Narration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participatory Video Intervention Group (Experimental): The Participatory Video intervention consists of 12 semi-structured, 2 hour group workshops over the course of a 6-month time period. Through facilitated discussion, participants will learn how to effectively work collaboratively as a member of the video production team. Together, they will choose what story of their shared experience with psychosis they would like to tell through documentary-video and how they plan to share it. Participants will be trained to operate all equipment required to bring their vision to life. Individuals will also have the opportunity, during the Participatory Video process, to create and share their own video clips, independent of the group, allowing participants to share their own video-narrative with others (friends, family members, public) as a means of engaging in dialogue around their personal experience with psychosis.
  Interventions: Behavioral: Participatory Video Intervention for Early Psychosis

INTERVENTIONS:
Behavioral: Participatory Video Intervention for Early Psychosis — The Participatory Video intervention consists of 12 semi-structured, 2 hour group workshops over the course of a 6-month time period. Through facilitated discussion, participants will learn how to effectively work collaboratively as a member of the video production team. Together, they will choose what story of their shared experience with psychosis they would like to tell through documentary-video and how they plan to share it. Participants will be trained to operate all equipment required to bring their vision to life. Individuals will also have the opportunity, during the Participatory Video process, to create and share their own video clips, independent of the group, allowing participants to share their own video-narrative with others (friends, family members, public) as a means of engaging in dialogue around their personal experience with psychosis.

SUMMARY:
Prior research has shown that people with psychotic illnesses, like schizophrenia, who make sense of and meaningfully integrate their psychotic experiences into their life story are more likely to recover from their illness. This process of developing a coherent narrative seems especially relevant for young people who are experiencing their first episode of psychosis. There is a need for interventions that can help facilitate the formation of recovery-oriented narratives, particularly in the early stage of illness. Participatory video is a group process that involves the facilitated creation of short documentary-style videos in which individuals are supported to reflect on and tell their personal stories. Although it has been used to foster self-identity, self-empowerment and "give voice" to a variety of marginalized and stigmatized populations, its use and evaluation as a clinical intervention has been limited.

The purpose of this study is to determine whether the novel use of participatory video facilitate narrative development and promote recovery for individuals with early psychosis is an effective, feasible, and acceptable means of treating youth in the early stages of psychotic illnesses. Although the current study is hypothesis generating in nature, the investigators are expecting that participating in the Participatory Video intervention will result in improvements in narrative development, symptoms, self-perceived recovery, self-esteem, self-stigma, social functioning and hope. Additionally, the investigators expect that Participatory Video intervention will prove to be acceptable to participants and a feasible intervention for early psychotic disorders.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a novel 12-session Participatory Video intervention, is an effective, feasible, and acceptable means of treating people in the early stages of psychotic illnesses.

We intend to randomly assign 20 patients being treated for psychotic illnesses in an early intervention program to a Participatory Video intervention group or treatment as usual group (control). Participants who are randomly assigned to the Participatory Video intervention will take part in 12 expert-facilitated group-based workshops over a period of 6 months, in which they will learn how to develop, film and produce a documentary-style video of their experiences with psychosis. At the end of the 12 workshops participants will have worked together to produce a group documentary video about their experiences with psychosis and, should they wish, individual videos about their own personal experiences with psychosis. Participants in the Participatory Video intervention group will receive the intervention in addition to any treatment they would usually receive through the early psychosis program. Those assigned to the treatment as usual group will continue to receive the standard care available to them in the early psychosis program.

Participants will be evaluated at baseline, at 6-months (immediately post-intervention) and at 9 months (3 months post-intervention) on a number measures. Participatory Video intervention acceptability will be assessed through the Client Satisfaction Questionnaire and qualitative interviews, feasibility will be assessed through recruitment, consent and completion rates, and efficacy will be assessed on measures of symptoms, functioning, subjective recovery, metacognitive capacity and narrative development.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be current outpatients of the Prevention and Early intervention Program for Psychoses (PEPP) at LHSC.
* PEPP only accepts patients with a first onset primary psychotic illness that have not been treated with an antipsychotic for longer than one month.
* Study participants must be within their first 3 years of being accepted into PEPP.
* Participants must be fluent in English, as determined by referring clinicians or researchers (in the case of advertisement referred participants) in order to meaningfully participate in the PV intervention and complete the assessment tools.

Exclusion Criteria:

* Potential participants that show high levels of disorganized or disruptive behaviour (as determined by a cut off score of 4 or 5 on the Positive Formal
* Thought Disorder or Bizarre Behaviour items of the Scale for the Assessment of Positive Symptoms [SAPS]) such that they will not be able to meaningfully participate in the MAC intervention will be excluded from the study.
* Participants must not be simultaneously participating in any other research projects involving active interventions at PEPP.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Scale for Assessment of Positive Symptoms (SAPS) | Baseline, Change from Baseline in SAPS at 6 months, change from baseline in SAPS at 9 months
Scale for Assessment of Negative Symptoms (SANS) | Baseline, Change from Baseline in SANS at 6 months, change from baseline in SANS at 9 months
Rosenberg Self-Esteem Schedule (RSES) | Baseline, Change from Baseline in RSES at 6 months, change from baseline in RSES at 9 months
Self-stigma of Mental Illness Scale (SSMIS) | Baseline, Change from Baseline in SSMIS at 6 months, change from baseline in SSMIS at 9 months
The Beck Hopelessness Scale (BHS) | Baseline, Change from Baseline in BHS at 6 months, change from baseline in BHS at 9 months
Maryland Assessment of Recovery in People with Serious Mental Illness Scale (MARS) | Baseline, Change from Baseline in MARS at 6 months, change from baseline in MARS at 9 months
Social Functioning Scale (SFS) | Baseline, Change from Baseline in SFS at 6 months, change from baseline in SFS at 9 months
Profile of Mood States (POMS) | Baseline, Change from Baseline in POMS at 6 months, change from baseline in POMS at 9 months
Client Satisfaction Questionnaire-8 | at 6 months (only to those in the Participatory Video Intervention Group)
Scale to Assess Narrative Development (STAND) | at 6 months
Metacognition Assessment Scale-Abbreviated (MAS-A) | at 6 months
Qualitative Focus Group - Participant descriptions of their experience with Participatory Video and suggestions for how to improve the Participatory Video intervention | at 6 months (only for those in the Participatory Video intervention group)
Individual Semi-Structured Interviews - Participant description of their individual experience with the PV intervention group and any changes they feel it may have engendered in their life | at 9 months (only for those in the Participatory Video-intervention group)
Recruitment Rates | baseline
Consent Rates | baseline
Completion Rates | at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Arlene MacDougall, M.Sc., M.D., Principal Investigator — London Health Sciences Centre/University of Western Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] France CM, Uhlin BD. Narrative as an outcome domain in psychosis. Psychol Psychother. 2006 Mar;79(Pt 1):53-67. doi: 10.1348/147608305X41001. PMID 16611421
- [Background] Roe D, Davidson L. Self and narrative in schizophrenia: time to author a new story. Med Humanit. 2005 Dec;31(2):89-94. doi: 10.1136/jmh.2005.000214. PMID 23674667
- [Background] Chadwick PK. Peer-professional first-person account: schizophrenia from the inside--phenomenology and the integration of causes and meanings. Schizophr Bull. 2007 Jan;33(1):166-73. doi: 10.1093/schbul/sbl034. Epub 2006 Sep 14. PMID 16973785
- [Background] Lysaker PH, Buck KD, Ringer J. The recovery of metacognitive capacity in schizophrenia across 32 months of individual psychotherapy: A case study. Psychotherapy Research 17(6): 713-720, 2007.
- [Background] Windell D, Norman RM. A qualitative analysis of influences on recovery following a first episode of psychosis. Int J Soc Psychiatry. 2013 Aug;59(5):493-500. doi: 10.1177/0020764012443751. Epub 2012 Apr 24. PMID 22532125
- [Background] McAdams DP, McLean KC. Narrative identity. Current Directions in Psychological Science 22(3): 233-238, 2013.
- [Background] Cavelti M, Kvrgic S, Beck EM, Rusch N, Vauth R. Self-stigma and its relationship with insight, demoralization, and clinical outcome among people with schizophrenia spectrum disorders. Compr Psychiatry. 2012 Jul;53(5):468-79. doi: 10.1016/j.comppsych.2011.08.001. Epub 2011 Sep 28. PMID 21956043
- [Background] Greben M, Schweitzer RD, Bargenquast R. Mechanisms of change in psychotherapy for people diagnosed with schizophrenia: the role of narrative reflexivity in promoting recovery. The Australian Journal of Rehabilitation Counselling 20(1): 1-14, 2014.
- [Background] Roe D, Hasson-Ohayon I, Mashiach-Eizenberg M, Derhy O, Lysaker PH, Yanos PT. Narrative enhancement and cognitive therapy (NECT) effectiveness: a quasi-experimental study. J Clin Psychol. 2014 Apr;70(4):303-12. doi: 10.1002/jclp.22050. Epub 2013 Oct 2. PMID 24114797
- [Background] White SA. (2003). Participatory video: Images that transform and empower. Sage.
- [Background] Yang KH. (2012). Reflexivity, participation, and video. The handbook of participatory video, 100-114.
- [Background] Shaw J, Robertson C. (1997). Participatory video: a practical approach to using video creatively in group development work. London (ua): Routledge.
- [Background] Bery R. (2003). Participatory video that empowers. Participatory video: Images that transform and empower, 102-121.
- [Background] Luttrell W, Restler V, Fontaine C. Youth Video-Making. Handbook of Participatory Video, 164, 2012.
- [Background] Norman CD, Yip AL. eHealth promotion and social innovation with youth: using social and visual media to engage diverse communities. Stud Health Technol Inform. 2012;172:54-70. PMID 22910502
- [Background] Lysaker PH, Ringer J, Maxwell C, McGuire A, Lecomte T. Personal narratives and recovery from schizophrenia. Schizophr Res. 2010 Aug;121(1-3):271-6. doi: 10.1016/j.schres.2010.03.003. Epub 2010 Mar 26. PMID 20347269
- See also: Cannabis and Psychosis — http://cannabisandpsychosis.ca/